CLINICAL TRIAL: NCT02216812
Title: Does Vitamin C Reduce Finger Stiffness After Distal Radius Fractures? A Placebo Randomized Controlled Trial
Brief Title: Does Vitamin C Reduce Finger Stiffness After Distal Radius Fractures?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Neal Chung-Jen Chen, Medical Doctor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2014P000561
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Results first posted 2018-09-17 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-08

CONDITIONS: Finger Stiffness; Distal Radius Fracture
Keywords: Finger stiffness; Range of motion; Distal radius fracture; Vitamin C
MeSH Terms: conditions — Wrist Fractures | interventions — Ascorbic Acid; WW Domain-Containing Oxidoreductase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 500 mg vitamin C (Experimental): Arm will take 1 pill of 500 mg vitamin C per day for 6 weeks
  Interventions: Drug: 500 mg vitamin c, 1 pill per day for 6 weeks
- Placebo (Placebo Comparator): Arm will take 1 placebo pill per day for 6 weeks
  Interventions: Drug: 1 placebo pill for 6 weeks

INTERVENTIONS:
Drug: 500 mg vitamin c, 1 pill per day for 6 weeks
  Arms: 500 mg vitamin C
Drug: 1 placebo pill for 6 weeks
  Arms: Placebo

SUMMARY:
The reported prevalence of disproportionate pain and disability among patients recovering from a fracture of the distal radius varies widely. Literature reports numbers between 1% and 37%, perhaps in part because it is poorly defined, known by so many different names, subjective, and unverifiable.

The investigators are interested in the effect of vitamin C after distal radius fractures on objective measurement of finger motion, patient reported outcome measures, and pain intensity, instead of the previously used, subjective and imprecise criteria for complex regional pain syndrome.

Patients presenting to the Hand and Orthopaedic Trauma Services of MGH with a distal radius fracture will be asked to participate in this clinical trial. Patient will be randomly assigned to take either placebo or vitamin C 500 mg until full finger motion is attained as regarded by the treating physician at follow-up or for 6 weeks.

The investigators hypothesize no difference in finger stiffness at 6 weeks measured by distance to palmar crease of the index through little finger between patients taking vitamin C or placebo after a distal radius fracture. Additionally, the investigators assess finger stiffness by range of motion and stiffness of the thumb, and difference in PROMIS upper extremity function and pain score both measured at six months.

ELIGIBILITY:
Inclusion Criteria:

* All adult (age 18 or greater) patients presenting to the Hand and Orthopaedic Trauma Services of the Massachusetts General Hospital (MGH) within two weeks of a fracture of the distal radius, either operatively or nonoperatively treated

Exclusion Criteria:

* Patients with severe kidney failure, known allergy for vitamin C or pregnancy
* Multiple fractures, except for ulna fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-12-22 (Actual); Study Completion 2017-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Chen, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 500 mg Vitamin C: Arm will take 1 pill of 500 mg vitamin C per day for 6 weeks
  500 mg vitamin c, 1 pill per day for 6 weeks
- Placebo: Arm will take 1 placebo pill per day for 6 weeks
  1 placebo pill for 6 weeks
Period: Overall Study
Arm/Group | 500 mg Vitamin C | Placebo
Started | 67 | 67
Completed | 57 | 62
Not Completed | 10 | 5
Not completed — Lost to Follow-up | 10 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 500 mg Vitamin C | Placebo | Total
Number analyzed (Participants) | 67 | 67 | 134
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48 (17) | 50 (17) | 49 (17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 52 | 99
  Male | 20 | 15 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-causcasian | 13 | 4 | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 67 | 67 | 134
Dominant extremity injured [Count of Participants; unit: Participants] — The number of participants whose injured arm is the same side as that of their dominant hand (i.e., the hand with which they write or perform fine motor skills).
  Participants | 32 | 32 | 64
Non-operative treatment [Count of Participants; unit: Participants] | 42 | 41 | 83
Carpal tunnel release [Count of Participants; unit: Participants] | 4 | 9 | 13
PROMIS Pain Interference CAT [Mean (Standard Deviation); unit: T-score] — The Patient Reported Outcome Information System (PROMIS) Pain Interference Computer Adaptive Test (CAT) is a computerized assessment measuring the amount pain interferes in the subjects' activities. It is scored using a T-score, and the average is 50 for the U.S. population. In a given PROMIS, a T scores above 50 represents more of the measured variable than the average. Investigators measured this at enrollment.
  T-score | 65 (6.4) | 61 (7.1) | 63 (7.0)

OUTCOME MEASURES:

1. Primary Outcome: Distance to Palmar Crease Index Through Small Finger
Description: To establish the distance to palmar crease, we asked patients to make a fist and determine the distance from nail tip to palmar crease for each individual digit using a ruler. We defined total distance to palmar crease as the sum of the values for the index, long, ring, and small fingers.
Time Frame: Day 1 (baseline), 6 weeks
Population: Some subjects were lost to follow up between enrollment, 6 week visit, and 6 month surveys.
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | 500 mg Vitamin C | Placebo
Number analyzed (Participants) | 67 | 67
Centimeters
  Day 1 (baseline) | 6.7 (6.7) | 7.1 (6.0)
  6 weeks: number analyzed (Participants) | 57 | 62
  6 weeks | 2.3 (4.0) | 2.0 (3.8)
Statistical Analysis 1: Comparison: 500 mg Vitamin C vs Placebo; We tested the null hypothesis that there is no difference in DPC six weeks after fracture of the distal radius between patients taking vitamin C and placebo; Test type: Other; p = 0.63, Regression, Linear

2. Secondary Outcome: Active Flexion Index Through Small Finger
Description: Active flexion will be measured using a handheld goniometer. We calculate total active flexion of the index through small finger by summing flexion at the metacarpo-phalangeal, proximal interphalangeal and distal interphalangeal joints
Time Frame: Day 1 (baseline), 6 weeks
Population: Some subjects were lost to follow up between enrollment, 6 week visit, and 6 month surveys.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | 500 mg Vitamin C | Placebo
Number analyzed (Participants) | 67 | 67
Degrees
  Day 1 (baseline) | 725 (159) | 732 (144)
  6 weeks: number analyzed (Participants) | 57 | 62
  6 weeks | 896 (108) | 904 (132)

3. Secondary Outcome: Thumb Motion
Description: Total active range of motion at the thumb combines active flexion at the metacarpo-phalangeal and interphalangeal joint, as well as palmar andabduction
Time Frame: Day 1 (baseline), 6 weeks
Population: Some subjects were lost to follow up between enrollment, 6 week visit, and 6 month surveys.
Measure: Mean (Standard Deviation); unit: Degrees
Arm/Group | 500 mg Vitamin C | Placebo
Number analyzed (Participants) | 67 | 67
Degrees
  Day 1 (baseline) | 161 (59) | 155 (49)
  6 weeks: number analyzed (Participants) | 57 | 62
  6 weeks | 229 (49) | 232 (46)

4. Secondary Outcome: PROMIS Upper Extremity - CAT
Description: The Patient Reported Outcome Information System (PROMIS) Upper Extremity Computer Adaptive Test (CAT) is a computerized assessment measuring the physical function of the upper extremity. It is scored using a T-score, and the average is 50 for the U.S. population. In a given PROMIS, a T-score above 50 represents more of the measured variable than the average. For this variable, a T-score above 50 indicates greater physical function than the average population.
Time Frame: Day 1 (baseline), 6 weeks, 6 months
Population: Some subjects were lost to follow up between enrollment, 6 week visit, and 6 month surveys.
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | 500 mg Vitamin C | Placebo
Number analyzed (Participants) | 67 | 67
T-score
  Day 1 (Baseline) | 26 (7.9) | 27 (7.5)
  6 weeks: number analyzed (Participants) | 57 | 62
  6 weeks | 35 (6.9) | 36 (8.4)
  6 months: number analyzed (Participants) | 48 | 50
  6 months | 48 (8.4) | 48 (9.1)

5. Secondary Outcome: 0-10 Ordinal Pain Score
Description: Measure Description: The Ordinal Pain Scale measures the amount of pain on a scale from 0, no pain, to 10, worst possible pain. The investigators will compare the change in pain between the two cohorts after 6 weeks of treatment and 6 months after treatment.
Time Frame: Day 1 (baseline), 6 weeks, 6 months
Population: Some subjects were lost to follow up between time of enrollment and 6 week and 6 month follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 500 mg Vitamin C | Placebo
Number analyzed (Participants) | 67 | 67
units on a scale
  Day 1 (baseline) | 3.5 (2.4) | 3.8 (2.6)
  6 weeks: number analyzed (Participants) | 57 | 67
  6 weeks | 1.6 (2.2) | 1.8 (1.9)
  6 months: number analyzed (Participants) | 48 | 50
  6 months | 1.4 (2.3) | 1.7 (2.2)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | 500 mg Vitamin C | Placebo
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/67
Other Adverse Events (participants affected / at risk) | 0/67 | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-22): https://cdn.clinicaltrials.gov/large-docs/12/NCT02216812/Prot_SAP_000.pdf